CLINICAL TRIAL: NCT04207099
Title: A 12-week, Prospective, Parallel Arm, Randomized Controlled Trial (RCT) Comparing Wound Area Reduction of Non-healing Diabetic Foot Ulcers With MolecuLight i:X Used in Standard of Care Compared to Standard of Care Alone
Brief Title: Comparing Wound Area Reduction of Non-healing DFUs Using MolecuLight i:X Versus Standard of Care
Acronym: WAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MolecuLight Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-014
Record Dates: First submitted 2019-11-29; First posted 2019-12-20 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Non Healing Diabetic Foot Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- ARM 1: Patients receive standard of care treatment for their diabetic foot ulcer
- ARM 2: Patients receive MolecuLight i:X guided treatment for their diabetic foot ulcer
  Interventions: Device: MolecuLight i:X Imaging Device

INTERVENTIONS:
Device: MolecuLight i:X Imaging Device — The MolecuLight i:X Imaging Device uses built-in light-emitting diodes (LEDs) emitting 405 nm violet excitation light to illuminate the wound during fluorescence imaging in (FL-Mode). The light excites biological components of the wound and surrounding tissues. Non-biological components may also fluoresce although their presence in wounds is less common, provided the wound has been cleaned following standard care protocols. The resulting wound fluorescence wavelengths emitted are typically between 420 - 700 nm in the visible wavelength spectrum. In FL-mode, a customized fluorescence emission filter, which is mechanically placed in front of the built in imaging sensor and allows real-time capture of wound, limits the visualization of fluorescence to wavelengths between 500-545 nm, which typically appears green in color, and 600-665 nm, which typically appears red in color.
  Groups: ARM 2

SUMMARY:
This is a 12 week, randomized controlled trial. There are 2 arms and 20 patients with non healing diabetic foot ulcer allocated in each arm. One arm receives i:X guided treatment and the other arm receives standard of care treatment. Our primary objective is to compare the wound area reduction in both arms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients presenting with chronic DFU
* The chronic DFU has a surface area that has reduced <25% in the previous 4 weeks1 prior to first study visit
* Patient has been receiving treatment for their DFU for less than 12 weeks.
* The chronic DFU is > 1 cm2 in area and less than 15 cm in length (max. diameter)
* 18 years or older
* Willing and able to make all required study visits

Exclusion Criteria:

* • Patients categorized as having a maintenance wound

  * Use of skin substitutes or hyperbaric oxygen therapy or surgical intervention
  * Treatment with an investigational drug within 1 month of enrolment
  * Presents with chronic (>10 mg/kg for >30 days) systemic corticoids before enrolment
  * Has ABI <0.5 (measured within 3 months of randomisation)
  * Undergoing chemotherapy or is immunocompromised
  * Diagnosed with Charcot disease or ulcers from electrical, chemical or radiation burns, or presents with collagen vascular disease, ulcer malignancy, untreated osteomyelitis or cellulitis
  * Recombinant or autologous growth factors or skin/dermal substitutes within 30 days of enrollment
  * Inability or unwillingness to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects presenting with non healing diabetic foot ulcer
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-02-14 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of change in wound area of diabetic foot ulcers in ARM 2 vs ARM 1 | 5 months
  ARM 2 vs ARM 1 Evaluate change in wound area over 12-week period

SECONDARY OUTCOMES:
Wound Healing Rate | 5 months
  ARM 1 vs. ARM 2
  1. Evaluate increase in wound healing rate over 12-week period
  2. Evaluate differences in clinical infection i. time to eradicate an infection ii. incidence of new infection (i.e. infection avoidance)
  3. Determine if MolecuLight i:X images taken at baseline can predict non-healing wounds, region for debridement and/or wounds at risk of infection (based on fluorescent signatures) at 6 and 12 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - ILD Research Centre, Vista, California
  - Northwell Comprehensive Wound Healing Center and Hyperbarics, Lake Success, New York

IPD SHARING:
Plan to Share IPD: Undecided